CLINICAL TRIAL: NCT05702034
Title: A Phase 3, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Demonstrate the Efficacy and Safety of Milvexian, an Oral Factor XIa Inhibitor, for Stroke Prevention After an Acute Ischemic Stroke or High-Risk Transient Ischemic Attack
Brief Title: A Study of Milvexian in Participants After an Acute Ischemic Stroke or High-Risk Transient Ischemic Attack- LIBREXIA-STROKE
Acronym: LIBREXIA-STROK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bristol Myers Squibb Company (BMS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR109231; 70033093STR3001 (Other: Janssen Research & Development, LLC); 2022-501176-26-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-01-19; First posted 2023-01-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke; Ischemic Attack, Transient
MeSH Terms: conditions — Ischemic Stroke | interventions — milvexian

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Milvexian (Experimental): Participants after an acute ischemic stroke or high-risk transient ischemic attack (TIA) who are receiving antiplatelet therapy standard-of-care (SAPT [single antiplatelet therapy] or DAPT [dual antiplatelet therapy]) will receive milvexian 25 milligrams (mg), orally, twice daily.
  Interventions: Drug: Milvexian
- Placebo (Placebo Comparator): Participants after an acute ischemic stroke or high-risk TIA who are receiving antiplatelet therapy standard-of-care (SAPT or DAPT) will receive placebo orally twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milvexian — Milvexian will be administered orally.
  Other Names: JNJ-70033093, BMS-986177
  Arms: Milvexian
Drug: Placebo — Placebo will be administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether milvexian compared to placebo reduce the risk of recurrent ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic Stroke: a neurological deficit attributable to an acute brain infarction and national institute of health stroke score scale (NIHSS) score less than or equal to (<=) 7 and at least 1 of the following: persistent signs or symptoms of the ischemic event at the time of randomization, or acute, ischemic brain lesion determined by standard-of-care neuroimaging, or participant underwent thrombolysis or thrombectomy, or transient ischemic attack (TIA): acute onset neurological deficit attributable to focal ischemia of the brain by history or examination, with complete symptom resolution of the deficit and no brain infarction on neuroimaging (example, computed tomography (CT) scan or magnetic resonance imaging (MRI), performed as part of standard medical practice), and ABCD2 Score greater than or equal to (>=) 6
* Participants will be randomized as soon as possible after determining eligibility and within 48 hours of onset of event.
* Current or planned antiplatelet treatment per international and/or local guidelines. If acetyl salicylic acid (ASA) is used, it will be limited to low dose (75 to 100 milligrams (mg)/day). Loading dose of antiplatelet agents (including ASA) are allowed per standard-of-care
* A female participant must agree not to be pregnant, breastfeeding, or planning to become pregnant until 4 days (5 half lives) after the last dose of study intervention
* Willing and able to adhere to the lifestyle restrictions specified in this protocol

Exclusion Criteria:

* Prior history of intracranial hemorrhage except subarachnoid hemorrhage greater than (>) 1 year prior with adequate treatment
* The index stroke or TIA is considered to have a cardio-embolic etiology based on local standard-of-care investigations and for which guidelines recommend anticoagulation
* The index stroke or TIA considered to have another known cause, not related to athero-thrombotic sources (treatment of acute stroke trial [TOAST] Other Determined Etiology), based on local standard-of-care investigations
* Increased risk of bleeding, including clinically significant bleeding within the previous 3 months or known bleeding diathesis or known activated partial thromboplastin time (aPTT) prolongation or spinal cord hemorrhage or retinal hemorrhage
* Current active liver disease, eg, acute hepatitis, known cirrhosis, including participants receiving antiviral treatment for hepatitis
* Known allergies, hypersensitivity, or intolerance to milvexian or its excipients

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Ischemic Stroke | Up to global targeted endpoint date (approximately 41 months)
  Time to first occurrence of ischemic stroke will be reported.

SECONDARY OUTCOMES:
Time to First Occurrence of any Component of the Composite of Cardiovascular Death (CVD), Myocardial Infraction (MI), or Ischemic Stroke | Up to global targeted endpoint date (approximately 41 months)
  Time to first occurrence of any component of the composite of CVD, MI, or ischemic stroke will be reported.
Time to First Occurrence of Ischemic Stroke | Up to Day 90
  Time to first occurrence of ischemic stroke in the first 90 days will be reported.
Time to First Occurrence of any Component of Major Adverse Vascular Events (MAVE) | Up to global targeted endpoint date (approximately 41 months)
  Time to first occurrence of any component of MAVE will be reported. MAVE is a composite of (CVD), myocardial infarction (MI), ischemic stroke, major adverse limb events (MALE), symptomatic pulmonary embolism (PE) or deep vein thrombosis (DVT).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (869):
- United States (122):
  - Banner Desert Medical Center, Mesa, Arizona
  - University of Arizona, Tucson, Arizona
  - Plaza Neuroscience Clinic, Fayetteville, Arkansas
  - Alta Bates Medical Center Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center - Cancer Center, Burbank, California
  - Mills Peninsula Health Services, Burlingame, California
  - Sutter Health - Eden Medical Center, Castro Valley, California
  - Neurology Center of North Orange County, Fullerton, California
  - Glendale Adventist Medical Center, Glendale, California
  - UC Irvine Healthcare Center, Irvine, California
  - Sharp Grossmont Hospital, La Mesa, California
  - Long Beach Memorial, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Mission Hospital Regional Medical Center, Mission Viejo, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Stanford Stroke Center, Palo Alto, California
  - Kaiser Permanente, Redwood City, California
  - University of California Davis Health System, Sacramento, California
  - Kaiser Permanente, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - Pacific Neuroscience Institute, Santa Monica, California
  - Harbor Ucla Medical Center, Torrance, California
  - Providence Little Company of Mary, Torrance, California
  - PIH Health Hospital, Whittier, California
  - University of Colorado, Aurora, Colorado
  - Nuvance Health Medical Practices Cardiology Danbury, Danbury, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Baptist Health, Miami, Florida
  - Advent Health Orlando, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Theia Clincial Research, LLC, Temple Terrace, Florida
  - Saint Marys Medical Center, West Palm Beach, Florida
  - Augusta University, Augusta, Georgia
  - Saint Alphonsus Regional Medical Center- Cancer Care Center, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Insight Hospital and Medical Center Chicago, Chicago, Illinois
  - Northshore University Healthsystem, Evanston, Illinois
  - St. Joseph's Regional Medical Center, Joliet, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Blessing Hospital, Quincy, Illinois
  - Javon Bea Hospital, Rockford, Illinois
  - Prairie Education And Research Cooperative, Springfield, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Community Hospital Cardiovascular Research, Munster, Indiana
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Ascension via Christi Research, Wichita, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Shady Grove Office, Rockville, Maryland
  - Comprehensive Neurology Services, Silver Spring, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - St John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Memorial Institute for Neurosciences and Multiple Sclerosis, Owosso, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Providence & Providence Park Hospital, Southfield, Michigan
  - M Health Fairview Ridges Hospital, Burnsville, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - University Of Minnesota Medical Center, Saint Louis Park, Minnesota
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - SSM Health DePaul Hospital, Bridgeton, Missouri
  - Cox Health, Springfield, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Capital Health Regional Medical Center, Trenton, New Jersey
  - Mercy Hospital, Buffalo, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - United Health Services, Johnson City, New York
  - Lenox Hill Hospital, Lake Success, New York
  - Long Island Jewish Med Ctr, New Hyde Park, New York
  - Weill Cornell Medical College, New York, New York
  - Lincoln Hospital, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Novant Health, Charlotte, North Carolina
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Summa Health System, Akron, Ohio
  - TriHealth Network, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Ascension Medical Group - St. John Clinic Infectious Disease, Tulsa, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St Vincent Medical Center, Portland, Oregon
  - Oregon Health And Science University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital Jeanes Campus, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Centennial Medical Center, Nashville, Tennessee
  - TriStar Skyline Medical Center, Nashville, Tennessee
  - Saint Thomas Health, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seton Medical Center, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - McGovern Medical School UT Physicians Neurosurgery Texas Medical Center, Houston, Texas
  - Houston Methodist Willowbrook Hospital, Houston, Texas
  - Emergency Medicine Covenant Medical Center, Lubbock, Texas
  - Sentara Medical Group, Norfolk, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Multiple Sclerosis Center at Evergreen, Kirkland, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - Mayo Clinic Health System, Eau Claire, Wisconsin
  - Mayo Clinic Health System, La Crosse, Wisconsin
- Argentina (22):
  - Fundacion Favaloro, Buenos Aires
  - Hospital Aleman, Buenos Aires
  - Sanatorio Finochietto, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Sanatorio Los Arcos, Buenos Aires
  - Sanatorio Guemes, CABA
  - Sanatorio Mater Dei, Ciudad Autonoma Buenos Aires
  - Hospital Gral Agudos Ignacio Pirovano, Ciudad Autonoma Buenos Aires
  - Clinica Adventista Belgrano, Ciudad Autonoma Buenos Aires
  - Hospital Municipal Dr Raul Alfredo Caccavo, Coronel Suárez
  - Clinica Privada Velez Sarsfield, Córdoba
  - Clínica Colombo, Córdoba
  - Hospital San Roque, Córdoba
  - Clínica Chutro, Córdoba
  - Sanatorio Allende, Córdoba
  - Sanatorio de la Canada, Córdoba
  - Hospital Cordoba, Córdoba
  - Hospital General de Agudos Dr. J. M. Ramos Mejia, Federal
  - Sanatorio Parque, Rosario
  - Hospital Interzonal General de Agudos Eva Perón, San Martín
  - Clinica Mayo de UMCB, San Miguel de Tucumán
  - Estudios Clinicos de los Arroyos, San Nicolás
- Australia (21):
  - Royal Adelaide Hospital, Adelaide
  - Flinders Medical Centre, Adelaide
  - Box Hill Hospital, Box Hill
  - Campbelltown Hospital, Campbelltown
  - Royal Prince Alfred Hospital, Camperdown
  - Monash Medical Centre, Clayton
  - St Vincent's Hospital - Melbourne, Fitzroy
  - Austin Health, Heidelberg
  - Royal Brisbane and Women's Hospital, Herston
  - Launceston General Hospital, Launceston
  - Liverpool Hospital, Liverpool
  - The Alfred Hospital, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - John Hunter Hospital, New Lambton Heights
  - Royal Melbourne Hospital, Parkville
  - Prince Of Wales Hospital, Randwick
  - Mater Hospital Brisbane, South Brisbane
  - Gold Coast University Hospital, Southport
  - Royal Darwin Hospital, Tiwi
  - Latrobe Regional Hospital, Traralgon
  - Princess Alexandra Hospital, Woolloongabba
- Austria (2):
  - Klinikum Klagenfurt am Worthersee, Klagenfurt
  - Klinikum Wels Grieskirchen, Wels
- Belgium (12):
  - ZNA Middelheim, Antwerp
  - Centre Hospitalier EPICURA Ath-Baudour-Hornu, Ath
  - Imeldaziekenhuis, Bonheiden
  - C.H.U. Brugmann, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - AZ Sint-Blasius, Dendermonde
  - UZA, Edegem
  - Az Groeninge, Kortrijk
  - Chu Tivoli, La Louvière
  - UZ Leuven, Leuven
  - CHC MontLegia, Liège
  - CHU Ambroise Pare, Mons
- Brazil (26):
  - Instituto das Pequenas Missionárias de Maria Imaculada - Hospital Madre Teresa, Belo Horizonte
  - Fundacao para o Desenvolvimento Medico Hospitalar (UNESP Botucatu), Botucatu
  - Hospital Brasilia, Brasília
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina da UNICAMP, Campinas
  - Hospital do Rocio, Campo Largo
  - Sociedade Literaria e Caritativa Santo Agostinho Hospital Sao Jose, Criciúma
  - Universidade Federal do Parana - Hospital de Clínicas, Curitiba
  - Instituto Presbiteriano Mackenzie - Hospital Universitario Evangelico Mackenzie, Curitiba
  - HGF - Hospital Geral de Fortaleza, Fortaleza
  - Associacao Hospital de Caridade Ijui, Ijuí
  - Clinica Neurologica e Neurocirurgica de Joinville, Joinville
  - Complexo Hospitalar de Niteroi, Niterói
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - IMV Pesquisa Neurológica, Porto Alegre
  - Associacao Educadora Sao Carlos AESC Hospital Mae De Deus, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Irmandade Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital Nove de Julho, São Paulo
  - Casa de Saude Santa Marcelina - Hospital Santa Marcelina, São Paulo
  - HC-UFTM - Hospital de Clínicas da Universidade Federal do Triângulo Mineiro, Uberaba
  - Hospital Estadual Central, Vitória
- Bulgaria (21):
  - Multiprofile Hospital for Active Treatment Puls, Blagoevgrad
  - MHAT Botevgrad EOOD, Botevgrad
  - MHAT Sveti Ivan Rilski, Dupnitsa
  - MHAT Sveti Ivan Rilski, Gorna Oryahovitsa
  - Multiprofile Hospital for Active Treatment - Haskovo, Haskovo
  - Mhat Sveti Georgi, Montana
  - MHAT - Pazardzhik AD, Pazardzhik
  - MHAT Avis - Medica OOD, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT Kaspela, Plovdiv
  - UMHAT Sveti Georgi, Plovdiv
  - UMHAT 'Kanev' EAD, Rousse
  - MHAT Southwest hospital OOD, Sandanski
  - MHAT Hadzhi Dimitar, Sliven
  - Medical Center St. Naum, Sofia
  - University First MHAT-Sofia St Joan Krastitel EAD, Sofia
  - Multiprofile Hospital For Active Treatment National Cardiology Hospital, Ead, Sofia
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - University Multiprofile Hospital for Active Treatment - Tsaritsa Yoanna - ISUL, EAD, Sofia
  - UMHATEM N I Pirogov, Sofia
  - University Multiprofile Hospital for Active Treatment- UMHAT Sveta Anna AD, Sofia
- Canada (19):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Lethbridge Regional Hospital, Lethbridge, Alberta
  - Medicine Hat Regional Hospital - Medical Arts Clinic, Medicine Hat, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Brandon Regional Health Centre, Brandon, Manitoba
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Trillium Health Partners, Mississauga, Ontario
  - Niagara Health System - Greater Niagara General Site, Niagara Falls, Ontario
  - Unity Health Toronto, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - CISSS de la Monteregie Centre, Greenfield Park, Quebec
  - CHU de Quebec - Hôpital de l' Enfant Jésus, Québec, Quebec
  - CHUS, Sherbrooke, Quebec
- Chile (4):
  - Hospital Base de Osorno, Osorno
  - Clinica Alemana de Santiago S.A., Santiago
  - Hospital Dipreca, Santiago
  - Hospital Clinico Vina del Mar, Viña del Mar
- China (78):
  - The People's Hospital of Anyang City, Anyang
  - Baoji Central Hospital, Baoji
  - Baogang Hospital, Inner Mongolia, Baotou
  - Xuanwu Hospital ,Capital Medical University, Beijing
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Jilin Province Peoples Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - Hunan Province People's Hospital The First Affiliated Hospital of Hunan Normal University, Changsha
  - The second Xiangya Hospital of Central South University, Changsha
  - Changsha Central Hospital, Changsha
  - Chengdu Second People's Hospital, Chengdu
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu
  - Chenzhou No.1 People's Hospital, Chenzhou
  - PLA Army Characteristic Medical Center, Chongqing
  - Affiliated Zhongshan Hospital of Dalian University, Dalian
  - Dalian Municipal Central Hospital, Dalian
  - Dazhou Central Hospital, Dazhou
  - People's Hospital of Deyang City, Deyang
  - Dongguan People s Hospital, Dongguan
  - Jiangxi Ganzhou Peoples Hospital, Ganzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Guangdong Second Provincial General Hospital, Guangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - Inner Mongolia People's Hospital, Hohhot
  - Qilu Hospital of Shandong University, Jinan
  - Shandong First medical university, Jinan
  - Jingdezhen No.1 People's Hospital, Jingdezhen
  - Shandong Jining No.1 People's Hospital, Jining
  - The No.2 Hospital affiliated to Guizhou Medical college, Kaili
  - First Peoples Hospital of Yunnan Province, Kunming
  - The First Hospital of Lanzhou University, Lanzhou
  - The Second People's Hospital of Lianyungang, Lianyungang
  - Liaocheng People s Hospital, Liaocheng
  - Linfen Central Hospital, Linfen
  - Linyi City People Hospital, Linyi
  - Liuzhou people's Hospital, Liuchow
  - No. 2 Hospital Affiliated to Henan Technical University, Luoyang
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Nanchong Central Hospital, Nanchong
  - Zhongda Hospital Southeast University, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Nanyang Central Hospital, Nanyang
  - Nanshi Hospital of Nanyang, Nanyang
  - Pingxiang People's Hospital, Pingxiang
  - Qingdao Municipal Hospital, Qingdao
  - The First Hospital of Qiqihar, Qiqihar
  - Shanghai Seventh People's Hospital, Shanghai
  - The First Affiliated Hospital of Shantou University Medical, Shantou
  - Shengjing Hospital Of China Medical University, Shenyang
  - The first people's hospital of Shenyang, Shenyang
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Second Affiliated Hospital of Soochow University, Suzhou
  - Tai An City Center Hospital, Taian
  - Shanxi Cardiovascular Hospital, Taiyuan
  - Shanxi Provincial People's Hospital, Taiyuan
  - Taizhou Peoples Hospital, Taizhou
  - Tianjin Medical University General Hospital, Tianjin
  - Tonghua Central Hospital, Tonghua
  - The first affiliated hospital of Xinjiang medical university, Ürümqi
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Ruian People's Hospital, Wenzhou
  - The Central Hospital of Wuhan, Wuhan
  - Wuxi 2nd Peoples Hospital, Wuxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Zhongshan Hospital, Xiamen University, Xiamen
  - Xiangtan Central Hospital, Xiangtan
  - Xuancheng People s Hospital, Xuancheng
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Affiliated Hospital of Yangzhou University, Yangzhou
  - Yanbian University Hospital, Yanji
  - Yantai Yuhuangding Hospital, Yantai
  - Yichang Central Pepole's Hospital, Yichang
  - Affiliated Hospital Of Guangdong Medical University, Zhanjiang
- Croatia (8):
  - Opca bolnica Bjelovar, Bjelovar
  - Clinic hospital Osijek, Osijek
  - Clinical Hospital Centre Rijeka, Rijeka
  - Clinical Hospital Center Split, Split
  - OB Varazdin, Varaždin
  - Clinical Hospital Centre Zagreb, Zagreb
  - Clinical Hospital Sestre Milosrdnice, Zagreb
  - University Hospital Sveti Duh, Zagreb
- Czechia (11):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Nemocnice Jihlava, Jihlava
  - Fakultni nemocnice Olomouc, Olomouc
  - Nemocnice AGEL Ostrava Vitkovice a s, Ostrava - Vitkovice
  - Nemocnice Pisek, a.s., Písek
  - Fakultni Nemocnice Ostrava, Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
  - Ustredni vojenske nemocnice Praha, Prague
- Denmark (6):
  - Ålborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus
  - Bispebjerg Og Frederiksberg Hospital, Copenhagen NV
  - Rigshospitalet, Glostrup Municipality
  - Herlev Hospital, Herlev
  - Herning Regional Hospital, Herning
- West Tallinn Central Hospital, Tallinn, Estonia
- Finland (3):
  - Helsinki University Hospital, HUS
  - Turun yliopistollinen keskussairaala, Turku
  - Vaasa Central Hospital, Vaasa
- France (26):
  - Centre Hospitalier du Pays d'Aix Service de Neurologie, Aix-en-Provence
  - CHRU Besancon Hopital Jean Minjoz, Besançon
  - Groupe Hospitalier Pellegrin CHU de Bordeaux, Bordeaux
  - CHU Bourg en Bresse, Bourg-en-Bresse
  - CHU de Brest - Hopital de la Cavale Blanche, Brest
  - Hopital Neurologique Pierre Wertheimer, Bron
  - Centre Hospitalier de Chartres, Chartres
  - CHU Clermont-Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital Raymond Poincare, Garches
  - Centre Hospitalier, La Roche-sur-Yon
  - CHR Metz Thionville Hopital de Mercy, Laquenexy
  - Hopital Roger Salengro - CHU Lille, Lille
  - CHU de Limoges Hopital Dupuytren, Limoges
  - Hopital de la Timone, Marseille
  - Centre Hospitalier Annecy Genevois, Metz-Tessy
  - Hopital Gui de Chauliac, Montpellier
  - Centre Hospitalier Universitaire de Nancy - Hôpital Central, Nancy
  - Hopital Lariboisiere, Paris
  - Hopital Saint Joseph, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Fondation Adolphe de Rothschild Hospital, Paris
  - Centre Hospitalier De Perpignan - Hopital Marechal Joffre, Perpignan
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - CHU Rouen Hopital Charles Nicolle, Rouen
  - Hopital Pierre Paul Riquet - Purpan, Toulouse
  - CHU Tours - Hopital Bretonneau - Maladies Infectieuses, Tours
- Germany (38):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Altenburger Land GmbH, Altenburg
  - Neurologische Klinik Bad Neustadt Saale, Bad Neustadt an der Saale
  - Vivantes Auguste Viktoria Klinikum, Berlin
  - Charite Campus Benjamin Franklin, Berlin
  - Vivantes Klinikum Neukoelln, Berlin
  - Vivantes Humboldt Klinikum, Berlin
  - Klinikum Dortmund gGmbH, Dortmund
  - Staedtisches Klinikum Dresden Standort Dresden Friedrichstadt, Dresden
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitatsklinikum Erlangen, Erlangen
  - Alfried Krupp Krankenhaus Ruettenscheid, Essen
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Frankfurt Goethe Universitaet, Frankfurt
  - Klinikum Frankfurt Hoechst GmbH, Frankfurt
  - Klinikum Friedrichshafen GmbH, Friedrichshafen
  - Philipps Universitaet Marburg Klinikum Fulda GAG, Fulda
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
  - Universitatsmedizin Gottingen, Göttingen
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Asklepios Klinik Wandsbeck, Hamburg
  - Asklepios Klinik Nord - Heidberg, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum Main Spessart, Lohr a. Main
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Medizinisches Zentrum Klinikum Lueneburg, Lüneburg
  - Johannes Wesling Klinikum Minden, Minden
  - Institut fuer Schlaganfall- und Demenzforschung, München
  - Universitaetsklinikum Muenster, Münster
  - Klinikum Ernst von Bergmann gGmbH, Potsdam
  - Nordwest Krankenhaus Sanderbusch, Sande
  - Helios Klinikum Schleswig, Schleswig
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (11):
  - Uni General Hospital of Alexandroupolis, Alexandroupoli
  - Laiko General Hospital of Athens, Athens
  - Alexandra General Hospital of Athens, Athens
  - General Hospital of Athens Attikon, Athens
  - Tzanio General Hospital of Piraeus, Athens
  - University General Hospital of Ioannina, Ioannina
  - University Hospital Of Larissa, Larissa
  - Ahepa University General Hospital of Thessaloniki, Thessaloniki
  - Hippokration Hospital, Thessaloniki
  - Papageorgiou General Hospital, Thessaloniki
  - G Papanikolaou Hospital of Thessaloniki, Thessaloniki
- Hong Kong (3):
  - The University of Hong Kong, Hong Kong
  - The Chinese University of Hong Kong, N T
  - North District Hospital, New Territories
- Hungary (16):
  - Péterfy Sándor utcai Kórház, Budapest
  - Semmelweis Egyetem, Budapest
  - Bajcsy-Zsilinszky Kórház és Rendelőintézet, Budapest
  - Esza-Kozep-budai Centrum, Uj Szent Janos Korhaz es Szakrendelo, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Orszagos Mentalis, Ideggyogyaszati es Idegsebeszeti Intezet, Budapest
  - Debreceni Egyetem Klinikai Központ,Infektológiai Klinika, Debrecen
  - Szent Pantaleon Kórház-Rendelointézet Dunaújváros, Dunaújváros
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Szent Damjan Gorogkatolikus Korhaz, Kisvárda
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Szent Lazar Megyei Korhaz, Salgótarján
  - Szent Borbala Hospital Tatabanya, Tatabánya
  - Javorszky Odon Korhaz, Vác
- India (52):
  - NHL Medical College (SVP Hospital IMSR), Ahmedabad
  - J L N Medical College and Attached Hospitals, Ajmer
  - Shree Krishna Hospital and Medical Research Center, Anand
  - Bangalore Medical College and Research Institute, Bangalore
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre (MRC), Belagavi
  - SUM Ultimate Medicare, Bhubaneswar
  - Apollo Hospitals, Bhubaneswar
  - S.P.Medical College & AG of Hospitals, Bikaner
  - Stanley Medical College, Chennai
  - Tamil Nadu Government Multi Super Speciality Hospital, Chennai
  - SIMS Multispecialty Hospital, Chennai
  - K.G. Hospital and PG Medical Institute, Coimbatore
  - ESIC Medical College and Hospital, Faridabad
  - Guru Gobind Singh Medical College and Hospital, Farīdkot
  - Institute of Neurological Sciences GNRC, Guwahati
  - Gauhati Medical College and Hospital, Guwahati
  - Paras Hospital, Gūrgaon
  - Nizams Institute of Medical Sciences, Hyderabad
  - Yashoda Super Speciality Hospitals, Hyderabad
  - Care Hospitals, Hyderbad
  - Shalby Hospital, Jaipur
  - Institute of Neurosciences Kolkata, Kolkata
  - Bangur Institute of Neurosciences and Psychiatry, Kolkata
  - Baby Memorial Hospital, Kozhikode
  - King Georges Medical University, Lucknow
  - Dayanand Medical College & Hospital, Tagore Nagar, Civil Lines, Ludhiana
  - Christian Medical College, Ludhiana
  - Mallikatta Neurocentre, Mangalore
  - B. Y. L. Nair Charitable Hospital & Topiwala National Medical College, Mumbai
  - Seth G S Medical College and KEM Hospital, Mumbai
  - JSS Hospital, Mysuru
  - Chopda Medicare & Research Centre, Nashik
  - Siddhi Hospital, Nashik
  - BLK Super Specialty Hospital, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Ruby Hall Clinic, Pune
  - Sahyadri Speciality Hospital, Pune
  - Synergy Superspeciality Hospital, Rajkot
  - All India Institute of Medical Sciences, Sumthāna
  - Institute of Neuroscience, Surat
  - Kiran Super Multispecialty Hospital, Surat
  - Bhaktivedanta Hospital & Research Institute, Thane
  - Government Medical College, Thiruvananthapuram
  - City Neurology Centre, Varanasi
  - Banaras Hindu University, Varanasi
  - Galaxy Life Care Services Pvt. Ltd, Varanasi
  - Christian Medical College, Vellore
  - Government Siddhartha Medical College, Vijayawada
  - King George Hospital, Visakhapatnam
  - Visakha Institute of Medical Sciences, Visakhapatnam
  - Government Medical College Vizianagaram, Vizianagaram
  - Mahatma Gandhi Memorial Hospital, Warangal
- Israel (9):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Health Corporation of Galilee Medical Center, Naharya
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Ziv Medical Center, Safed
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (24):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia Presidio Spedali Civili, Brescia
  - Azienda Ospedaliera Istituti Ospitalieri di Cremona, Cremona
  - Nuovo Ospedale San Giovanni Battista, Foligno
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Azienda Sanitaria Locale 1 Umbria - Ospedale di Gubbio e Gualdo Tadino, Gubbio
  - Ospedale Vito Fazzi, Lecce
  - Azienda Ospedaliera della Provincia di Lecco_Presidio Ospedaliero 'A. Manzoni' - S.C.di Cardiologia, Lecco
  - Ospedale San Salvatore, L’Aquila
  - Ospedale Apuane, Massa
  - Ospedale San Raffaele, Milan
  - Nuovo Ospedale Civile S.Agostino - Estense, Modena
  - Fondazione Istituto Neurologico Casimiro Mondino, Pavia
  - Azienda Unita Sanitaria Locale Umbria 1 Ospedale di Citta di Castello, Perugia
  - Azienda Ospedaliera di Perugia Ospedale S.Maria della Misericordia, Perugia
  - Azienda Ospedaliera Ospedale Santa Corona, Pietra Ligure
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Arcispedale S Maria Nuova (Civic Hospital), Reggio Emilia
  - Ospedale S. Eugenio, Roma
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Policlinico Umberto I, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda sanitaria universitaria Giuliano Isontina ASU GI, Trieste
  - ASUI Santa Maria della Misericordia di Udine, Udine
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (70):
  - Funabashi Municipal Medical Center, Chiba
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Steel Memorial Yawata Hospital, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Saiseikai Fukuoka General Hospital, Fukuoka
  - Fukuoka Neurosurgical Hospital, Fukuoka
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Japanese Red Cross Takayama Hospital, Gifu
  - Tokai University Hachioji Hospital, Hachiōji
  - Seirei Hamamatsu General Hospital, Hamamatsu
  - JA Hiroshima General Hospital, Hatsukaichi
  - Saitama Medical University International Medical Center, Hidaka
  - Higashihiroshima Medical Center, Higashihiroshima-shi
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji-shi
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hiroshima City Asa Citizens Hospital, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima
  - Ja Toride Medical Center, Ibaraki
  - Ina Central Hospital, Ina-shi
  - National Hospital Organization Kanazawa Medical Center, Ishikawa
  - National Hospital Organization Kagoshima Medical Center, Kagoshima
  - Fukuoka Tokushukai Hospital, Kasuga-shi
  - Nagoya Tokushukai General Hospital, Kasugai-shi
  - St Marianna University Hospital, Kawasaki
  - Kokura Memorial Hospital, Kitakyushu-shi
  - Hospital of the University of Occupational and Enviromental Health, Kitakyushu-shi
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Fukuoka Higashi Medical Center, Koga
  - Asama Nanroku Komoro Medical Center, Komoro-shi
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Chugoku Rosai Hospital, Kure
  - Shinkoga Clinic, Kurume-shi
  - Koseikai Takeda Hospital, Kyoto
  - Kyoto University Hospital, Kyoto
  - Maebashi Red Cross Hospital, Maebashi
  - Matsubara Tokushukai Hospital, Matsubara-shi
  - Nagasaki University Hospital, Nagasaki
  - NHO Nagoya Medical Center, Nagoya
  - Hyogo Medical University Hospital, Nishinomiya Shi
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - Omuta City Hospital, Omuta-Shi
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Osaka University Hospital, Osaka
  - Rinku General Medical Center, Osaka
  - Jinikai Makita General Hospital, Ōta-ku
  - Saga University Hospital, Saga
  - Kyoyukai Sainokuni Higashi Omiya Medical Center, Saitama-shi
  - Ijinkai Nakamura Memorial Hospital, Sapporo
  - Sendai City Hospital, Sendai
  - Kohnan Hospital, Sendai
  - Shimonoseki City Hospital, Shimonoseki-shi
  - Kanmon Medical Center, Shimonoseki-shi
  - Jichi Medical University Hospital, Shimotsuke
  - Keio University Hospital, Shinjuku-ku
  - Shizuoka City Shizuoka Hospital, Shizuoka Aoi-ku
  - National Cerebral and Cardiovascular Center, Suita-Shi
  - Nippon Medical School Hospital, Tokyo
  - NTT Medical Center Tokyo, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
  - Kyorin University Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - National Hospital Organization Toyohashi Medical Center, Toyohasi-shi
  - Toyota Memorial Hospital, Toyota-shi
  - University of Tsukuba Hospital, Tsukuba
  - Juntendo University Hospital Urayasu, Urayasu-shi
  - Uwajima City Hospital, Uwajima-shi
  - Sanyudo Hospital, Yonezawa-shi
- Latvia (2):
  - Riga East Clinical University Hospital, Riga
  - Pauls Stradins Clinical University Hospital, Riga
- Lithuania (2):
  - Vilnius University Hospital Santariskiu Clinic, Public Institution, Vilnius
  - Republican Vilnius University Hospital, Public Institution, Vilnius
- Malaysia (8):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Tengku Ampuan Rahimah, Klang
  - Hospital University Sains Malaysia, Kota Bharu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Kebangsaan Malaysia Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
  - Hospital Seberang Jaya, Seberang Jaya
  - Hospital Sungai Buloh, Sungai Buloh
- Mexico (6):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez, Distrito Federal
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Centro de Investigacion Clinica Chapultepec S.A. de C.V., Morelia
  - PRISMA Neurociencias A.C., San Luis Potosí City
- Netherlands (3):
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Bernhoven Uden, Uden
- New Zealand (6):
  - Auckland City Hospital, Auckland
  - Hawkes Bay Hospital, Hastings
  - Middlemore Hospital, Otahuhu
  - Rotorua Hospital, Rotorua
  - Tauranga Hospital, Tauranga
  - Wellington Hospital, Wellington
- Philippines (14):
  - Cebu Doctors University Hospital, Cebu
  - Davao Doctors Hospital, Davao City
  - St.Paul's Hospital-Iloilo, Iloilo City
  - West Visayas State University Medical Center, Iloilo City
  - Mary Mediatrix Medical Center, Lipa City
  - Manila Doctors Hospital, Manila
  - Chinese General Hospital & Medical Center, Manila
  - Metropolitan Medical Center, Manila
  - Amang Rodriguez Memorial Medical Center, Marikina City
  - San Juan de Dios Educational Foundation, Inc (Hospital), Pasay
  - The Medical City, Pasig
  - St. Luke's Medical Center, Quezon
  - Capitol Medical Center Inc., Quezon City
  - GreenCity Medical Center, San Fernando City
- Poland (21):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital Sw Lukasza w Boleslawcu Centrum Profilaktyki I leczenia udarow Mozgu, Bolesławiec
  - Szpital Uniwersytecki NR 1 IM Dr Antoniego Jurasza, Bydgoszcz
  - Samodzielny Publiczny Wojewodzki Szpital Specjalistyczny w Chelmie, Chelmie
  - Samodzielny Publiczny ZOZ w Dzialdowie, Działdowo
  - SP Specjalistyczny Szpital Zachodni im. Jana Pawla II, Grodzisk Mazowiecki
  - Samodzielny Publiczny Zespol Zakladow Opieki Zdrowotnej Medicam Gryfice, Gryfice
  - Uniwersyteckie Centrum Kliniczne im prof K Gibinskiego SUM, Katowice
  - SPSK nr 7 SUM w Katowicach Gornoslaskie Centrum Medyczne im Prof Leszka Gieca, Katowice Ochojec
  - Oddzial Ortopedii i Traumatologii Narzadu Ruchu Szpital Specjalistyczny im Ludwika Rydygiera, Krakow
  - Wojewodzki Szpital Zespolony w Lesznie Oddzial Neurologiczny z Pododzialem udarowym, Leszno
  - Uniwersytecki Szpital Kliniczny nr 1 im. N. Barlickiego, Lodz
  - III Szpital Miejski im. Dr. K. Jonschera w Lodzi, Lodz
  - 1 Wojskowy Szpital Kliniczny Z Poliklinika SPZOZ W Lublinie, Lublin
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Wojewodzki Szpital Specjalistyczny nr 3 w Rybniku, Rybnik
  - Zespol Opieki Zdrowotnej w Skarzysku-Kamiennej Szpital Powiatowy im. M.Curie-Sklodowskiej, Skarżysko-Kamienna
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Specjalistyczny Szpital Miejski im. M.Kopernika, Torun
  - Uniwersyteckie Centrum Kliniczne, Warsaw
  - Szpital Specjalistyczny im. F. Ceynowy Szpitale Pomorskie, Wejherowo
- Portugal (12):
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitário de Coimbra - Hospitais da Universidade de Coimbra, Coimbra
  - Centro Hospitalar Cova da Beira, E.P.E., Covilha
  - Uls Alto Ave - Hosp. Sra. Da Oliveira Guimaraes, Guimarães
  - Centro Hospitalar de Lisboa Central, Lisbon
  - Uls Lisboa Ocidental - Hosp. Egas Moniz, Lisbon
  - Centro Hospitalar de Lisboa Norte Hospital Santa Maria, Lisbon
  - H. Santo António - Centro Hospitalar do Porto, Porto
  - Hospital Garcia de Orta, EPE, Pragal
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E, Santa Maria da Feira
  - Centro Hospitalar de Vila Nova de Gaia Espinho E P E, Vila Nova de Gaia
  - Centro Hospitalar de Trás-os-Montes e Alto Douro, EPE - Unidade de Vila Real, Vila Real
- Romania (6):
  - Spitalul Clinic Judetean de Urgenta Arad, Arad
  - Spitalul de Psihiatrie si Neurologie Brasov, Brasov
  - Institutul National de Neurologie si Boli Neurovasculare Bucuresti, Bucharest
  - Emergency Clinical County Hospital Constanta, Constanța
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Pius Brinzeu, Timișoara
- Serbia (8):
  - Special Hospital for Cerebrovascular Disease Sveti Sava, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
  - Clinical Center of Vojvodina, Novi Sad
  - General Hospital 'Dr Radivoj Simonovic', Sombor
  - Health Center Subotica, Subotica
  - General Hospital Uzice, Užice
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Neuroscience Institute, Singapore
- Slovakia (13):
  - FNsP F. D. Roosevelta Banska Bystrica, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Bratislava
  - Univerzitna nemocnica L. Pasteura Kosice, Košice
  - Nemocnica AGEL Levice, s.r.o., Levice
  - Nemocnica S Poliklinikou SV. Barbory, Lučenec
  - Univerzitná nemocnica Martin, Martin
  - Fakultna nemocnica s poliklinikou Nove Zamky, Nové Zámky
  - Centrum Intervencnej Neuroradiologie a Endovaskularnej Liecby CINRE, Petržalka
  - Nemocnica s poliklinikou Spisska Nova Ves, a.s., Spišská Nová Ves
  - Nemocnica Trebisov, Trebišov
  - FN Trencin, Trenčín
  - Fakultna nemocnica Trnava, Trnava
  - Fakultna nemocnica s poliklinikou v Ziline, Žilina
- South Africa (10):
  - Iatros International, Bloemfontein
  - Tread Research, Cape Town
  - Naidoo A, Durban
  - Synergy Biomed Research Institute (SBRI), East London
  - TASK Central, George
  - Garda, RA, Johannesburg
  - Into Research, Pretoria
  - Dr J.M. Engelbrecht Trial Site, Somerset West
  - Drs Sarvan and Moodley, Tongaat
  - Clinical Projects Research SA (PTY) LTD, Worcester
- South Korea (32):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Pusan National University Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Chosun university hospital, Gwangju
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Catholic Kwandong University International ST Marys Hospital, Incheon
  - Jeju National University Hospital, Jeju Special
  - Chungnam National University Hospital, Sejong-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Hanyang University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Seoul National University Boramae Hospital, Seoul
  - Ewha Woman's University Seoul Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Soon Chun Hyang Univ.Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Uijeongbu Eulji Medical Center Eulji University, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - Yongin Severance Hospital, Yongin-si
- Spain (32):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Gral. de Albacete, Albacete
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp. Del Mar, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. Dr. Josep Trueta, Girona
  - Hosp. Univ. de Bellvitge, L'Hospitalet de Llobregat
  - Hosp. Univ. Arnau de Vilanova de Lleida, Lleida
  - Complejo Hosp Ruber Juan Bravo, Madrid
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. de La Paz, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Puerta Del Sur, Móstoles
  - Hosp. Univ. Son Espases, Palma de Mallorca
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. Virgen Del Rocio, Seville
  - Hosp Univ de Tarragona Joan Xxiii, Tarragona
  - Hosp. Mutua Terrassa, Terrassa
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. Clinico Univ. de Valladolid, Valladolid
  - Hosp. Alvaro Cunqueiro, Vigo
  - Hosp. Univ. Miguel Servet, Zaragoza
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Hässleholms sjukhus, Hässleholm
  - Skanes universitetssjukhus, Malmo
  - Skaraborgs sjukhus Skövde, Skövde
- Switzerland (5):
  - Kantonsspital Aarau, Aarau
  - Universitatsspital Basel, Basel
  - Inselspital Universitatsspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Kantonsspital St Gallen, Sankt Gallen
- Taiwan (14):
  - Changhua Christian Hospital, Changhua
  - Chia-Yi Christian Hospital, Chia-Yi City
  - Chang Gung Memorial Hospital, Chiayi Branch, Chiayi City
  - National Taiwan University Hospital, Douliu
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Keelung
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - En Chu Kong Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital- Linkou, Taoyuan
- Thailand (8):
  - Phramongkutklao Hospital and Medical College, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkoknoi
  - Maharaj Nakorn Chiang Mai hospital Faculty of Medicine, Chiang Mai
  - Lampang Hospital, Muang
  - Srinagarind Hospital, Nai Mueang Subdistrict Mueang
  - King Chulalongkorn Memorial Hospital, Pathum Wan
  - Prasat Neurological Institute, Rajathevi
- Turkey (Türkiye) (17):
  - Ankara University, Ankara
  - Hacettepe Universitesi Hastanesi, Ankara
  - Gazi University Medical Faculty, Ankara
  - Bursa Yuksek Ihtisas Training and Research Hospital, Bursa
  - Dicle University Medical Faculty, Diyarbakır
  - Firat University Hospital, Elâzığ
  - Erciyes University Medical Faculty, Erciyes
  - Bakirkoy Prof. Dr. Mazhar Osman Mental Health and Neurology Hospital, Istanbul
  - Bakirkoy Training and Research Hospital, Istanbul
  - Sisli Etfal Research Training Hospital, Istanbul
  - Kartal Dr Lutfi Kirdar Egitim ve Arastirma Hastanesi, Istanbul
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Medical Faculty, Izmir
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Sakarya University Training and Research Hospital, Sakarya
  - Ondokuz Mayis University, Samsun
  - Izmir Katip Celebi University Ataturk Training and Research Hospital, Turkey
- United Kingdom (29):
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospital Monklands, Airdrie
  - Royal United Hospital, Bath
  - Bury Care Organisation, Bury
  - Cheltenham General Hospital, Cheltenham
  - Darent Valley Hospital, Dartford
  - Doncaster Royal Infirmary, Doncaster
  - Ninewells Hospital, Dundee
  - Hairmyres Hospital, East Kilbride
  - Royal Devon and Exeter Hospital(Wonford), Exeter
  - Queen Elizabeth University Hospital, Glasgow
  - Calderdale Royal Hospital, Halifax
  - Hull Royal Infirmary, Hull
  - Leicester General Hospital, Leicester
  - Lincoln County Hospital, Lincoln
  - Royal London Hospital, London
  - Kings College Hospital, London
  - Luton and Dunstable Hospital, Luton
  - Arrowe Park Hospital, Metropolitan Borough of Wirral
  - Nottingham University Hospitals, Nottingham
  - Derriford Hospital, Plymouth
  - Royal Preston Hospital, Preston
  - Royal Hallamshire Hospital, Sheffield
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Musgrove Park Hospital, Taunton
  - Royal Cornwall Hospital, Truro
  - Pinderfields General Hospital - Dept. of Neurology, Wakefield
  - Watford General Hospital, Watford
  - York Hospital, York
- Vietnam (9):
  - Da Nang General Hospital, Da Nang
  - Bach Mai Hospital, Hanoi
  - 103 Military Hospital, Hanoi
  - Hanoi Medical University Hospital, Hanoi
  - People's Hospital 115, Ho Chi Minh City
  - Thong Nhat HOSPITAL, Ho Chi Minh City
  - University Medical Center Ho Chi Minh city, Ho Chi Minh City
  - Gia Dinh People Hospital, Ho Chi Minh City
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency